CLINICAL TRIAL: NCT02859324
Title: A Phase 1/2, MultiCenter, Open-label, Dose Finding Study to Assess the Safety, Tolerability and Preliminary Efficacy of CC-122 in Combination With Nivolumab in Subjects With Unresectable Hepatocellullar Carcinoma (HCC) Following First Line Treatment Failure
Brief Title: A Safety and Efficacy Study of CC-122 in Combination With Nivolumab in Subjects With Unresectable Hepatocellular Carcinoma (HCC)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-122-HCC-002; 2016-000112-15 (EudraCT Number)
Record Dates: First submitted 2016-08-04; First posted 2016-08-09 (Estimated); Results first posted 2021-05-11 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-04

CONDITIONS: Carcinoma, Hepatocellular
Keywords: CC-122; Nivolumab; Hepatocellular Carcinoma; Phase 1/2; Safety
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — 3-(5-amino-2-methyl-4-oxoquinazolin-3(4H)-yl)piperidine-2,6-dione; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CC-122 with Nivolumab (Experimental): CC-122 orally 5/7 days with nivolumab Intravenously (IV) 3mg/kg every 2 weeks. Cohorts of up to 6 subjects per dose level until Recommended Phase 2 dose (RP2D).
  Interventions: Drug: CC-122; Drug: Nivolumab

INTERVENTIONS:
Drug: CC-122
Drug: Nivolumab

SUMMARY:
CC-122-HCC-002 is a Phase 1/2 dose escalation and expansion clinical study of CC-122 in combination with nivolumab in subjects with unresectable hepatocellular carcinoma (HCC) who have progressed after or were intolerant to no more than 2 previous systemic therapies for unresectable HCC, or are naïve to systemic therapy.

DETAILED DESCRIPTION:
Study population included subjects who had progressed after or were intolerant to no more than 2 previous systemic therapies for unresectable HCC, or are naïve to systemic therapy.

The dose escalation part of the study was designed to explore three dose levels of CC-122 to identify the recommended phase 2 dose (RP2D) to be used in the expansion phase. Approximately 20 subjects were to be enrolled in the dose escalation part of the study. Subjects could be treated for up to 2 years, or until progression of disease, unacceptable toxicity, subject/physician decision, withdrawal of consent, death. Safety follow up until 28 days after CC122 treatment and 90 days after nivolumab treatment. RECIST 1.1 criteria was used to determine response. Survival follow up until death, withdrawal of consent, or the study closes. Subjects were permitted to continue treatment beyond progression (TBP) if they continue to meet protocol criteria, had stable performance status, had clinical benefit, other treatment options were discussed. A separate ICF was signed to continue TBP.

During the dose escalation phase, CC-122 was administered orally 5 consecutive days out of 7 (5 days on/2 days off weekly) on Days 1 to 5, 8 to 12, 15 to 19 and 22 to 26 of each 28-day cycle. Once the RP2D for dosing of CC-122 in combination with nivolumab was defined, expansion (Phase 2) would start. A modified 3+3 dose escalation design was used to identify the initial toxicity of the combination. Up to six subjects were concurrently enrolled into a dose level. Decisions as to which dose level to enroll a new subject were based on the number of subjects enrolled and evaluable, the number of subjects experiencing DLTs, and the number of subjects enrolled but who are not yet evaluable for toxicity in the current cohort at the time of new subject entry. A Safety Review Committee (SRC) comprised of investigators participating in the study made dose escalation decisions based on these criteria.

After completion of the Dose Escalation Phase, the Dose Expansion Phase of the study did not proceed due to the changing landscape in the treatment of HCC. There were no additional safety concerns or safety signals identified in the dose escalation phase of the study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must satisfy the following criteria to be enrolled in the study:
* Subject is ≥ 18 years of age at the time of signing the informed consent form (ICF)
* Subject has a confirmed pathologic diagnosis of Hepatocellular carcinoma (HCC) according to the American Association for the Study of Liver Diseases (AASLD) Guidelines.
* Subjects who have progressed after or were intolerant to no more than 2 previous systemic therapies for unresectable HCC, or are naïve to systemic therapy.
* Subject has at least one measurable lesion according to RECIST 1.1.
* Subject has a life expectancy of ≥ 12 weeks
* Subject has an Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 or 1
* Subject has adequate hematologic function and adequate hepatic function at screening

Exclusion Criteria:

* The presence of any of the following will exclude a subject from enrollment:
* Subject has received more than 2 previous systemic therapies for Hepatocellular carcinoma (HCC).
* Subject has received previous treatment with any anti-PD-1 (Programmed death 1) or anti-PD-L1 (PD-1 ligand receptor) antibody

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-09-20 (Actual); Primary Completion 2020-03-27 (Actual); Study Completion 2020-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Akshay Patel, Study Director — Celgene Corporation
Locations (14):
- United States (4):
  - UCLA Division of Hematology Oncology, Los Angeles, California
  - University of Florida, Gainesville, Florida
  - NYU Langone Medical Center, New York, New York
  - Mary Crowley Cancer Research, Dallas, Texas
- France (4):
  - Institut Paoli Calmettes, Marseille
  - Centre Eugene Marquis, Rennes
  - Institut Universitaire du Cancer IUCT - Oncopole, Toulouse
  - Institut Gustave Roussy Hematologie, Villejuif
- Italy (3):
  - IRCCS - Istituo Clinico Humanitas - Humanitas Cancer Center, Milan
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Istituto Nazionale Tumori Regina Elena, Roma
- Spain (3):
  - Hospital Universitario Vall D Hebron, Barcelona
  - Hospital Ramon y Cajal, Madrid
  - Hospital 12 de Octubre, Madrid

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 21 participants treated
Groups:
- CC-122 2mg + Nivolumab: CC-122 2.0 mg orally 5 consecutive days out of 7 (5 days on/2 days off weekly) on Days 1 to 5, 8 to 12, 15 to 19 and 22 to 26 of each 28-day cycle, and nivolumab 3.0 mg/kg intravenously (IV) every 2 weeks.
- CC-122 3mg + Nivolumab: CC-122 3.0 mg orally 5 consecutive days out of 7 (5 days on/2 days off weekly) on Days 1 to 5, 8 to 12, 15 to 19 and 22 to 26 of each 28-day cycle, and nivolumab 3.0 mg/kg intravenously (IV) every 2 weeks.
- CC-122 4mg + Nivolumab: CC-122 4.0 mg orally 5 consecutive days out of 7 (5 days on/2 days off weekly) on Days 1 to 5, 8 to 12, 15 to 19 and 22 to 26 of each 28-day cycle, and nivolumab 3.0 mg/kg intravenously (IV) every 2 weeks.
Period: Overall Study
Arm/Group | CC-122 2mg + Nivolumab | CC-122 3mg + Nivolumab | CC-122 4mg + Nivolumab
Started | 7 | 9 | 5
Completed (Completed = Did not discontinue study) | 0 | 0 | 0
Not Completed | 7 | 9 | 5
Not completed — Death | 4 | 6 | 5
Not completed — Other reasons | 3 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CC-122 2mg + Nivolumab | CC-122 3mg + Nivolumab | CC-122 4mg + Nivolumab | Total
Number analyzed (Participants) | 7 | 9 | 5 | 21
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.9 (10.32) | 60.4 (11.75) | 66.4 (10.06) | 63.0 (10.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1 | 2
  Male | 7 | 8 | 4 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 3 | 5 | 12
  Unknown or Not Reported | 3 | 6 | 0 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 0 | 1 | 0 | 1
  White | 4 | 2 | 5 | 11
  Not collected or reported | 3 | 6 | 0 | 9

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Dose Limiting Toxicities (DLTs)
Description: During dose escalation, the DLT assessment period is defined as Days 1 to 28 of Cycle 1 including the predose assessments specified for Day 1 of Cycle 2.
  A DLT is defined as any of the following toxicities occurring within the DLT assessment window unless the event can clearly be determined to be unrelated to the drug.
Time Frame: 28 days
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | CC-122 2mg + Nivolumab | CC-122 3mg + Nivolumab | CC-122 4mg + Nivolumab
Number analyzed (Participants) | 7 | 9 | 5
Participants | 1 | 1 | 2

2. Primary Outcome: Incidence and Severity of Treatment-Emergent Adverse Events (TEAEs)
Description: During dose escalation, the TEAE phase 1 assessment period is defined as Days 1 to 28 of Cycle 1 including the predose assessments specified for Day 1 of Cycle 2.
  Number of participants who experienced a TEAE during the course of the study.
Time Frame: From first dose up to 28 days (CC-122) or 90 days (nivolumab) post-last dose (up to 2 years)
Population: All treated participants
Measure: Number; unit: Number of participants
Arm/Group | CC-122 2mg + Nivolumab | CC-122 3mg + Nivolumab | CC-122 4mg + Nivolumab
Number analyzed (Participants) | 7 | 9 | 5
Number of participants
  TEAEs | 7 | 9 | 5
  Participants with Grade 3-4 TEAEs | 7 | 6 | 4
  Participants with Grade 5 TEAEs | 2 | 0 | 3
  Participants with serious TEAEs | 6 | 5 | 4
  Participants with TEAE leading to discontinuation of CC-122 | 2 | 1 | 3
  Participants with TEAE leading to discontinuation of nivolumab | 1 | 1 | 3
  Participants with TEAE leading to discontinuation of both study drugs | 1 | 1 | 2

3. Primary Outcome: Objective Response Rate (ORR) by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Description: ORR is is defined as the number and percentage of participants with a best overall response (BOR) of confirmed complete response (CR) or partial response (PR).
Time Frame: up to 2 years
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | CC-122 2mg + Nivolumab | CC-122 3mg + Nivolumab | CC-122 4mg + Nivolumab
Number analyzed (Participants) | 7 | 9 | 5
Percentage of participants | 42.9 [9.9 to 81.6] | 0 [0.0 to 33.6] | 0 [0.0 to 52.2]

4. Secondary Outcome: Disease Control Rate (DCR) by RECIST 1.1
Description: DCR is is defined as the number and percentage of participants with a best overall response (BOR) of confirmed complete response (CR) or partial response (PR) or stable disease (SD).
Time Frame: up to 2 years
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | CC-122 2mg + Nivolumab | CC-122 3mg + Nivolumab | CC-122 4mg + Nivolumab
Number analyzed (Participants) | 7 | 9 | 5
Percentage of participants | 71.4 [29.0 to 96.3] | 44.4 [13.7 to 78.8] | 80.0 [28.4 to 99.5]

5. Secondary Outcome: Duration of Response (DoR) by RECIST 1.1
Description: Duration of response is measured from the date the criterion is first met for CR/PR using RECIST 1.1 rules (whichever is first recorded) until the first date when progressive disease using RECIST 1.1 is documented or death occurred.
Time Frame: up to 2 years
Population: All treated participants
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | CC-122 2mg + Nivolumab | CC-122 3mg + Nivolumab | CC-122 4mg + Nivolumab
Number analyzed (Participants) | 7 | 9 | 5
Days | NA [NA to NA] — Median not reached as insufficient progression events among responders | NA [NA to NA] — Median not reached as insufficient progression events among responders | NA [NA to NA] — Median not reached as insufficient progression events among responders

6. Secondary Outcome: Progression-Free Survival (PFS) by RECIST 1.1
Description: Progression-Free Survival (PFS) is defined as the time from the first dose date of study drug until tumor progression or death, whichever occurs first. A subject who has neither progressed nor died or who progresses or dies after an extended lost-to-follow up time (two or more missed assessments) is censored on the date of last adequate tumor assessment. Subjects without valid baseline or post-baseline tumor assessments are censored on their first dose date.
  Median and the 2-sided 95% confidence interval (CI) are based on Kaplan-Meier estimate of progression-free survival and time to progression using both observed and censored data.
Time Frame: up to 2 years
Population: All treated participants
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | CC-122 2mg + Nivolumab | CC-122 3mg + Nivolumab | CC-122 4mg + Nivolumab
Number analyzed (Participants) | 7 | 9 | 5
Days | 130.0 [42.0 to NA] — Upper limit not calculable as upper CI bound does not cross 50% threshold | 95.0 [51.0 to 144.0] | 122.0 [56.0 to 166.0]

7. Secondary Outcome: Overall Survival (OS) by RECIST 1.1
Description: Overall Survival (OS) is measured as the time from the first dose of study drug to death from any cause. Participants who have no death reported are censored at the last contact date the participant is known to be alive.
  Median and the 2-sided 95% confidence interval (CI) are based on Kaplan-Meier estimate of progression-free survival and time to progression using both observed and censored data.
Time Frame: up to 2 years
Population: All treated participants
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | CC-122 2mg + Nivolumab | CC-122 3mg + Nivolumab | CC-122 4mg + Nivolumab
Number analyzed (Participants) | 7 | 9 | 5
Days | 320.0 [96.0 to NA] — Upper limit not calculable as upper CI bound does not cross 50% threshold | 303.0 [196.0 to NA] — Upper limit not calculable as upper CI bound does not cross 50% threshold | 135.0 [95.0 to 387.0]

8. Secondary Outcome: Time to Progression (TTP) by RECIST 1.1
Description: Time to Progression (TTP) is defined as the time from the first dose date of study drug until tumor progression; TTP does not include death. The censoring rules are the same as PFS except that deaths without progression are censored at last adequate tumor assessment.
  Median and the 2-sided 95% confidence interval (CI) are based on Kaplan-Meier estimate of progression-free survival and time to progression using both observed and censored data.
Time Frame: up to 2 years
Population: All treated participants
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | CC-122 2mg + Nivolumab | CC-122 3mg + Nivolumab | CC-122 4mg + Nivolumab
Number analyzed (Participants) | 7 | 9 | 5
Days | NA [42.0 to NA] — Median not reached as insufficient progression events among responders | 95.0 [51.0 to 144.0] | 166.0 [56.0 to 166.0]

9. Secondary Outcome: Maximum Observed Concentration (Cmax)
Description: Blood was collected according to intensive and sparse sampling strategies to estimate the population pharmacokinetic (PK) of CC-122 when administered in combination with nivolumab.
Time Frame: 28 days
Population: Pharmacokinetic (PK) Evaluable Population -All participants who enrolled and received at least one dose of either investigational product (IP) and had at least one measurable concentration of CC-122 or nivolumab.
  Note: Nivolumab participants did not qualify for data analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | CC-122 2mg + Nivolumab | CC-122 3mg + Nivolumab | CC-122 4mg + Nivolumab
Number analyzed (Participants) | 2 | 9 | 1
ng/mL | 56.3 (48.4) | 81.0 (32.8) | 82.6 (NA) — Only 1 participant

10. Secondary Outcome: Area Under the Concentration Time Curve (AUC)
Description: as for outcome 9
Time Frame: 28 days
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | CC-122 2mg + Nivolumab | CC-122 3mg + Nivolumab | CC-122 4mg + Nivolumab
Number analyzed (Participants) | 2 | 9 | 1
h*ng/mL | 235.3 (17.3) | 399.8 (29.7) | 257.9 (NA) — Only 1 participant

11. Secondary Outcome: Time to Maximum Concentration (Tmax)
Description: as for outcome 9
Time Frame: 28 days
Population: as for outcome 9
Measure: Median (Full Range); unit: hour
Arm/Group | CC-122 2mg + Nivolumab | CC-122 3mg + Nivolumab | CC-122 4mg + Nivolumab
Number analyzed (Participants) | 2 | 9 | 1
hour | 0.5 [0.5 to 0.5] | 1.0 [0.5 to 2.0] | 1.0 [1.0 to 1.0]

12. Secondary Outcome: Terminal Half-life (T-HALF)
Description: as for outcome 9
Time Frame: 28 days
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | CC-122 2mg + Nivolumab | CC-122 3mg + Nivolumab | CC-122 4mg + Nivolumab
Number analyzed (Participants) | 2 | 8 | 0
hour | 8.4 (61.4) | 6.4 (42.1) |

13. Secondary Outcome: Apparent Volume of Distribution (Vz/F)
Description: as for outcome 9
Time Frame: 28 days
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter
Arm/Group | CC-122 2mg + Nivolumab | CC-122 3mg + Nivolumab | CC-122 4mg + Nivolumab
Number analyzed (Participants) | 0 | 1 | 0
liter |  | 40.1 (NA) — Only 1 participant value |

ADVERSE EVENTS:
Time Frame: From first dose up to 28 days (CC-122) or 90 days (nivolumab) post-last dose (up to 2 years) for all serious and non-serious adverse events. For all-cause mortality, the timeframe of reporting is over the entirety of the study (ca. 3.5 years).
Arm/Group | CC-122 2mg + Nivolumab | CC-122 3mg + Nivolumab | CC-122 4mg + Nivolumab
All-Cause Mortality (participants affected / at risk) | 4/7 | 6/9 | 5/5
Serious Adverse Events (participants affected / at risk) | 6/7 | 5/9 | 4/5
Other Adverse Events (participants affected / at risk) | 7/7 | 9/9 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CC-122 2mg + Nivolumab (N=7) | CC-122 3mg + Nivolumab (N=9) | CC-122 4mg + Nivolumab (N=5)
Ascites (Gastrointestinal disorders) | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Disease progression (General disorders) | 1 | 0 | 0
General physical health deterioration (General disorders) | 1 | 0 | 2
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0 | 0
Abdominal wall abscess (Infections and infestations) | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0
Liver abscess (Infections and infestations) | 0 | 0 | 1
Peritonitis bacterial (Infections and infestations) | 1 | 0 | 0
Pulmonary sepsis (Infections and infestations) | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CC-122 2mg + Nivolumab (N=7) | CC-122 3mg + Nivolumab (N=9) | CC-122 4mg + Nivolumab (N=5)
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 1
Neutropenia (Blood and lymphatic system disorders) | 2 | 5 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 2 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 0
Eye pain (Eye disorders) | 0 | 0 | 1
Eyelid rash (Eye disorders) | 0 | 1 | 0
Lacrimation increased (Eye disorders) | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 3 | 1 | 0
Ascites (Gastrointestinal disorders) | 2 | 1 | 2
Constipation (Gastrointestinal disorders) | 2 | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 4 | 1
Asthenia (General disorders) | 4 | 1 | 1
Chills (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 3 | 2
General physical health deterioration (General disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 1 | 4 | 2
Pyrexia (General disorders) | 1 | 2 | 2
Swelling (General disorders) | 1 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 2 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 2 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 2 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Tinea versicolour (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 1 | 3
Amylase increased (Investigations) | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 4
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 2 | 0 | 2
Blood creatine increased (Investigations) | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1
Blood phosphorus decreased (Investigations) | 1 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0
Lipase increased (Investigations) | 2 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 1
Troponin I increased (Investigations) | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Torticollis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Aphasia (Nervous system disorders) | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 0
Lacunar infarction (Nervous system disorders) | 0 | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0
Anxiety disorder (Psychiatric disorders) | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Exfoliative rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hair colour changes (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 2 | 3
Hypertension (Vascular disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2017-08-29): https://cdn.clinicaltrials.gov/large-docs/24/NCT02859324/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-30): https://cdn.clinicaltrials.gov/large-docs/24/NCT02859324/SAP_001.pdf